CLINICAL TRIAL: NCT05510011
Title: Clinical and Radiological Outcomes of Composite Tibial and Femoral Allograft and Tantalum Cone Reconstructions in Total Knee Replacement Revision
Brief Title: Allograft and Tantalum Cone Reconstruction in TKA Revision
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL22_0013
Record Dates: First submitted 2022-01-25; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-01

CONDITIONS: Tantalum; Bone Loss; Allograft
Keywords: Tantalum; Allograft; TKA revision using tantalum cone and/or allograft
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A new surgical technique of reconstruction for bone loss in TKA revision using tantalum cone and allograft.

Study of radiological and clinical outcomes.

ELIGIBILITY:
Inclusion criteria:

* > 18 years old
* TKA revision using tantalum cone or allograft

Exclusion criteria:

* <18 years old
* no reconstruction used in TKA revision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women attending for 3rd timester scan
Sampling Method: Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-02-20 (Estimated); Study Completion 2023-02-21 (Estimated)

PRIMARY OUTCOMES:
Rate of Survivorship of the implant | day 1
  Survivorship of the implant

CONTACTS AND LOCATIONS:
Overall Officials: Louis DAGNEAUX, PHU, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC